CLINICAL TRIAL: NCT02489812
Title: Music Distraction Strategy in Children Dental Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Junia Maria Serra-Negra, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UFMG
Record Dates: First submitted 2015-06-26; First posted 2015-07-03 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Children Behavior
Keywords: children; behavior; anxiety; dentistry
MeSH Terms: conditions — Behavior; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- music (Experimental): The Mozart Symphony No 40 in G minor K550 was played in headphones. While the child received restorative treatment in the teeth she heard music in a session and was subjected to other dental treatment session without listening to music. The cardiac and respiratory frequencies were measured with children's finger oximeter while the child listened to music and also in session in which she did not hear music. Changes in the measurements obtained by the oximeter showed levels of anxiety.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — This cross over trial aimed to analyze the use of music as a distraction resource during children dental treatment, evaluating their cardiac and respiratory frequency. Thirty-four children took part in this study, 16 boys and 18 girls, from 4 to 6 years old, with no previous dental experience, who had two carious lesions on occlusal surfaces of molars,
  Other Names: The Mozart Symphony No 40 in G minor K550

SUMMARY:
Music plays an important role reassuring helping reduce anxiety. Anxiety can be an interference factor in promoting oral health for children with high levels of anxiety tend to have negative behavior at the dentist. High oxygen levels and heart and respiratory frequencies are associated with high levels of anxiety. The objective of this study was to test the use of music in decreased cardiac and respiratory frequency of treated patients listening to music and being treated without hearing music.

DETAILED DESCRIPTION:
Feelings like anxiety can alter the levels of blood oxygenation from individuals in different situations, like during dental treatment. This cross over trial aimed to analyze the use of music as a distraction resource during children dental treatment, evaluating their cardiac and respiratory frequency. Thirty-four children took part in this study, 16 boys and 18 girls, from 4 to 6 years old, with no previous dental experience, who had two carious lesions on occlusal surfaces of molars, from the 2 municipalities of southeast Brasil. Children were selected through oral clinical exams, conducted in public schools. After parents signed a written consent; children were allocated in two groups: treatment with music (G1) and treatment without music (G2). Children acted as controls of themselves: the cross between groups allowed all children to be treated with and without music. Three dental visits were, scheduled in a weekly basis, the first for anamnesis and clinical examination; the second and third for the modified atraumatic restorative treatment (ARTm). The Mozart Symphony No 40 in G minor K550 was played in headphones. Cardiac and respiratory frequencies were obtained using a pulse oximeter, with the measures being taken in three moments: in the beginning of the treatment, during the intervention (use of a rotating device) and at the end of the treatment. Data were compiled and analyzed through the statistic software Statistical Analyse. The Wilcoxon test was used for inter and intra groups comparison (p<0,050).

Music worked as a reassuring instrument during children dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Without children experience provided at the dentist
* Healthy children and without syndromes
* Children with normal hearing
* Children with two occlusal carious lesions with loss of enamel and dentin to 2/3 wherever possible to carry out the treatment technique Atraumatic Restorative adapted.

Exclusion Criteria:

* Children with syndromes
* Children without normal hearing
* Children thal not collaborated with the dentist
* Children with hospital and/or dental experience

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of participants | 3 months
  Children were selected through oral clinical exams, conducted in public schools.

SECONDARY OUTCOMES:
Composite measure of Cardiac and respiratory frequencies using a pulse oximeter | 6 months